CLINICAL TRIAL: NCT06789640
Title: Impact of Vitamin C Supplementation on the Hospital Outcomes in Children Undergoing Corrective Heart Surgery for Congenital Heart Diseases
Brief Title: Impact of Vitamin C Supplementation on Hospital Outcomes in Children Undergoing Corrective Heart Surgery for Congenital Heart Diseases
Acronym: RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hoda Atef Abdelsattar Ibrahim, Hoda Atef Abdelsattar Ibrahim, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MS-588-2023; MS-588-2023 (Other: MS-588-2023)
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Congenital Heart Disease (CHD)
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional (Experimental): Vitamin C will be given before admission in the immediate preoperative preceding 7 days (the dose 30 -45 mg per day ) in oral drops preparations
  Inflammatory markers including CRP , TLC ,PNI , GPS NLR will be checked on admission and on discharge and compared between cases and controls Hospital length stay will also be compared between the two groups
  Interventions: Other: Vitamin C
- The control group (Placebo Comparator): A placebo will be given before admission in the immediate preoperative preceding 7 days (the dose 30 -45 mg per day ) in oral drops preparations
  Inflammatory markers including CRP , TLC ,PNI , GPS NLR will be checked on admission and on discharge and compared between cases and controls Hospital length stay will also be compared between the two groups
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Vitamin C — Vitamin C will be given before admission in the immediate preoperative preceding 7 days (the dose 30 -45 mg per day ) in oral drops preparations
  Inflammatory markers including CRP , TLC ,PNI , GPS NLR will be checked on admission and on discharge and compared between cases and controls Hospital length stay will also be compared between the two groups
  Arms: Interventional
Other: Placebo — Placebo will be given before admission in the immediate preoperative preceding 7 days (the dose 30 -45 mg per day ) in oral drops preparations
  Inflammatory markers including CRP , TLC ,PNI , GPS NLR will be checked on admission and on discharge and compared between cases and controls
  Arms: The control group

SUMMARY:
Vitamin C will be given before admission in the immediate preoperative preceding 7 days (the dose 30 -45 mg per day ) in oral drops preparations

Inflammatory markers including CRP , TLC ,PNI , GPS NLR will be checked on admission and on discharge and compared between cases and controls Hospital length stay will also be compared between the two groups

ELIGIBILITY:
Inclusion Criteria:

* Children in the first two years who will be for corrective surgery for heart diseases congenital heart diseases
* Pediatric patients whose parents or caregivers agree to be enrolled in the study.
* Risk Adjustment for Congenital Heart Surgery -1 (RACHS-1) for Evaluation of Mortality in Children Undergoing Cardiac Surgery : the first two categories (Thiagarajan and C. Laussen 2015)

Exclusion Criteria:

* Pediatric patients with associated comorbid conditions.

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-02-19 (Estimated); Primary Completion 2025-04-19 (Estimated); Study Completion 2025-04-19 (Estimated)

PRIMARY OUTCOMES:
The improvemnents of Ejection Fraction between the two groups | 7-10 days
  Each group wil be evaluated for the eiection fraction before and after the operation and the improvement will be compared

IPD SHARING:
Plan to Share IPD: Undecided